CLINICAL TRIAL: NCT02909049
Title: Open Randomized Clinical Trial to Examine Individual Pain Tolerance in the Use of Two Anesthetic Techniques to Perform Saturation Prostate Biopsy
Brief Title: Clinical Trial to Examine Individual Pain Tolerance in the Use of Two Anesthetic Techniques to Perform Saturation Prostate Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Principal Investigator, José Luis Ponce Díaz-Reixa, MD, Complexo Hospitalario Universitario de A Coruña
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO - CHUAC - BPSat - 001.
Record Dates: First submitted 2016-04-19; First posted 2016-09-21 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Prostatic Cancer
Keywords: Prostate Biopsy; Local Anesthesia; Pain; Biopsy of prostate
MeSH Terms: conditions — Prostatic Neoplasms; Pain | interventions — Midazolam; Mepivacaine; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTROL (Active Comparator): Saturation prostate biopsy under intravenous sedation MIDAZOLAM 1,5 mg per kilogram intravenous, 5 minutes prior to biopsy FENTANILE 0,05 mg per kilogram intravenous, 3 minutes prior to biopsy KETAMINE 0.5 mg per kilogram intravenous, 1 minute prior to biopsy
  Interventions: Drug: MIDAZOLAM; Drug: FENTANILE; Drug: KETAMINE
- EXPERIMENTAL (Experimental): Saturation prostate biopsy under local anesthesia MEPIVACAÍNE 2% 10 millimeters periprostatic block at base and ápex, bilaterally.
  Interventions: Drug: MEPIVACAÍNE

INTERVENTIONS:
Drug: MIDAZOLAM — Intravenous bolus anesthesia 5 minutes previous to saturation prostate biopsy.
  Other Names: MIDAZOLAM 15mg/3ml ATC N05CD08 MAN 65319
  Arms: CONTROL
Drug: MEPIVACAÍNE — Local periprostatic anesthesia infiltration, previous to saturation prostate biopsy.
  Other Names: MEPIVACAINE 2% ATC N01BB03 MAN 62606
  Arms: EXPERIMENTAL
Drug: FENTANILE — Intravenous bolus anesthesia 3 minutes previous to saturation prostate biopsy.
  Other Names: FENTANILE 0,05 mg/ml ATC N01AH01 MAN 41764
  Arms: CONTROL
Drug: KETAMINE — Intravenous bolus anesthesia 1 minute previous to saturation prostate biopsy.
  Other Names: KETAMINE 50 mg/ml ATC N01AX03 Marketing Authorisation number 47034
  Arms: CONTROL

SUMMARY:
To assess the effectiveness of two anesthetic techniques by measuring the pain through visual analog scale (VAS), to obtain saturation prostate biopsies.

DETAILED DESCRIPTION:
To assess the effectiveness of two anesthetic techniques by measuring the pain through visual analog scale (VAS), to obtain saturation prostate biopsies.

Anesthetic technique (control) - Intravenous sedation with Midazolam, Fentanile and Ketamine.

Anesthetic technique (intervention) - Regional Mepivacaine infiltration of periprostatic region.

ELIGIBILITY:
Inclusion Criteria:

* Male patient
* Persistence of suspected prostate cancer by altering the prostatic specific antigen and / or digital rectal examination.
* Two previous negative prostate biopsies .
* Age < 75 years.
* Signature of informed consent to perform prostate biopsy.
* Signature of informed consent for the study.

Exclusion Criteria:

* Age > 75 years.
* Absence of consent or refusal to the study .
* Presence of prostate cancer in previous biopsy observation .
* Medical-surgical patient's problems, absolutely contraindicating biopsy under local anesthesia.
* Presence of any allergies to medications involved in the study .
* Patient's clinical situation that does not allow an outpatient operation and aftercare required .
* Medical condition of the patient, preventing the realization of outpatient biopsy.
* No companion.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04; Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Change in visual analog scale (VAS) | 1 hour baseline
  Change in visual analog scale (VAS) from baseline and after prostate biopsy

SECONDARY OUTCOMES:
Number of patients with complications after anesthesic procedure and prostate biopsy procedure, after 24 hours of the procedure and at end of study visit. All units will be measured as numbers. | One week
  To assess the safety of the procedure and complications in the use of each of the anesthetic techniques during saturation prostate biopsy. Safety events will be measured during saturation prostate biopsy and after recovery, during 24 hours. Number of patients with complications after anesthesic procedure and prostate biopsy procedure. Number of patients with complications after 24 hours of the procedure. Number of patients with complications at end of study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Ponce, MD, Principal Investigator — Complejo Hospitalario Universitario, A Coruña
Locations (1):
- Jose Luis Ponce Diaz-Reixa, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No